CLINICAL TRIAL: NCT05750641
Title: The Efficacy of Removal of Animal Milk From the Diet in Functional Dyspepsia: A Cross-sectional Study
Status: Completed | Type: Observational
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Sponsor
Other Study IDs: Functional Dyspepsia and Milk
Record Dates: First submitted 2023-02-20; First posted 2023-03-02 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-02

CONDITIONS: Dyspepsia; Gastrointestinal System Disease
Keywords: functional dyspepsia; milk; dairy products
MeSH Terms: conditions — Dyspepsia; Digestive System Diseases | interventions — Guidelines as Topic

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- diet group: those who removed milk and dairy products under the advice of a dietician without medical treatment.
  Interventions: Other: removing milk and dairy products from diets without medical treatment
- free-diet group: According to current standard algorithms and guidelines, appropriate treatment for FD types was arranged for the patient group who preferred to receive a free diet.
  Interventions: Other: According to current standard algorithms and guidelines, appropriate treatment for FD types.

INTERVENTIONS:
Other: removing milk and dairy products from diets without medical treatment — A specialist dietician prepared a diet list based on providing adequate balanced nutrition and is handed over to the diet group without any medical treatment
  Groups: diet group
Other: According to current standard algorithms and guidelines, appropriate treatment for FD types. — According to current standard algorithms and guidelines, appropriate treatment for FD types was arranged for the patient group who preferred to receive a free diet
  Groups: free-diet group

SUMMARY:
The goal of this observational study is to learn about compare the effect of removing animal milk from diets on the symptoms of FD patients in describe participant population.

The main question it aims to answer are:

• Can removing milk and dairy from diets be used to treat FD patients?

The participants will be divided into two groups and will do the following;

* removing milk and dairy products under the advice of a dietician without medical treatment
* receiving medical treatment without restricted diet.

Researchers will compare two groups to the effect of removing milk from diet on the symptoms of FD patients.

DETAILED DESCRIPTION:
In this cross-sectional cohort study, 120 patients with FD diagnosed by the Rome IV criteria were included. Patients were divided equally into two groups; those who removed milk and dairy products under the advice of a dietician without medical treatment and those who did not. For determining the severity of symptoms, "The gastrointestinal Symptom Rating Scale (GSRS)" was used at the onset of the study and the end of the one-month follow-up period.

Between the two groups, there was no statistically significant difference regarding age, body mass index (BMI), frequency and duration of symptoms, weight changes in the last six months, FD subtypes, and upper GI endoscopy results (p>0.05). Female patients outnumbered men in the animal milk removal group (p=0.01). Although the patients in the animal milk removal group had higher GSRS scores at the beginning (p=0.01), both groups had similar GSRS scores at the end of the study (p=0.99). After one month follow-up period, GSRS scores have improved in both groups compared to the baseline (p=0.01). However, the decrease in the GSRS total symptom score was significantly higher in the animal milk removal group compared to the free diet group (p=0.01). In the evaluation of GSRS symptom subsets, a statistically higher reduction was observed in 7 of the 15 subsets in the animal milk removal group compared to the free-diet group (p<0.05).

Of the 120 FD patients who followed up for one month, 60 who removed milk products had a more significant reduction in GSRS symptom score and 7 of the 15 symptom subset scores than 60 patients receiving an unrestricted diet.

ELIGIBILITY:
Inclusion Criteria:

* between the ages of 18-65
* having at least one of the complaints of postprandial fullness, early satiety, epigastric burning and pain
* the onset of the complaint is at least 6 months ago and at least one complaint has been going on at least 3 days a week for the last 3 months
* no underlying organic pathology is detected in the examinations.

Exclusion Criteria:

* being outside the age range of 18-65
* having alarm symptoms such as vomiting, gastrointestinal bleeding, and weight loss of 5% or more in the last 3 months
* presence of comorbidities such as dementia, CVD, psychiatric diseases
* covid-19 positivity during the research

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients between the ages of 18-65 admitted to the gastroenterology outpatient clinic between September 2020 and March 2021, fulfilling the Rome IV Consensus criteria for the diagnosis of FD, were included in the study in a cross-sectional and prospective manner according to the order of admission
Sampling Method: Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
The comparing the scores of symptom subsets of the two patient groups | one month
  Gastrointestinal Symptom Rating Scale

CONTACTS AND LOCATIONS:
Locations (1):
- Bezmialem Vakif Univercity, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
The transfer of individual participant data in the study to electronic media was not provided.